CLINICAL TRIAL: NCT00876330
Title: CERT-HIT: A Multimodal Intervention to Improve Antihypertensive and Lipid-lowering Therapy
Brief Title: Improving Antihypertensive and Lipid-Lowering Therapy
Acronym: CERT2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven Simon, Site Principal Investigator, VA Boston Healthcare System
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1U18HS016970-01 (AHRQ)
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Hyperlipidemia; Hypertension
Keywords: Clinical Decision Support Systems; Hyperlipidemia; Hypertension
MeSH Terms: conditions — Hyperlipidemias; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Receives Hypertension and Hyperlipidemia Intervention using Clinical Decision Support.
  Interventions: Other: Clinical Decision Support for Hypertension; Other: Automated Telephone Outreach for Antihypertensive Therapy
- 2 (Experimental): Receives Hypertension and Hyperlipidemia Intervention with automated telephone outreach.
  Interventions: Other: Clinical Decision Support for Lipid-lowering Therapy; Other: Automated Telephone Outreach for Lipid-lowering Therapy

INTERVENTIONS:
Other: Clinical Decision Support for Hypertension — Clinical decision support alerts for antihypertensive therapy
  Arms: 1
Other: Automated Telephone Outreach for Antihypertensive Therapy — Automated Telephone Outreach to patients for antihypertensive medication therapy.
  Arms: 1
Other: Clinical Decision Support for Lipid-lowering Therapy — Clinical Decision Support alerts for Lipid-lowering medication therapy.
  Arms: 2
Other: Automated Telephone Outreach for Lipid-lowering Therapy — Automated telephone outreach to patients for Lipid-lowering medication therapy.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the impact of electronic health record clinical decision support and automated telephone outreach on antihypertensive and lipid-lowering therapy in ambulatory care.

DETAILED DESCRIPTION:
The quality of care delivered in physicians' offices is suboptimal. Underuse of proven, potentially life-saving medications, such as anti-hypertensive agents and statins for lipid-lowering, is unfortunately no exception. Data from more than 70 million people collected for the 2005 HEDIS Report Card show that fewer than half of those patients at high risk for myocardial infarction have adequately controlled lipids and fewer than 70% of patients with hypertension have blood pressure controlled; annually this suboptimal treatment accounts for more than 10,000 avoidable deaths, $333 million in avoidable hospital costs, 27.2 million sick days and $4.5 billion in lost productivity.

The "care-gaps" in the management of blood pressure and lipids arise from numerous barriers to optimal practice at the level of the system, the provider, and the patient. Process evaluations of quality improvement efforts have cited several barriers as the most important: inadequate time, resources, and support; limitations in computer technology, including insufficient information management; little use of formal change processes; too many competing priorities; a lack of agreement about the desired changes; and inadequate physician engagement.

Both computerized clinical decision support (CDS) in the context of a robust electronic health record (EHR) and automated telephone outreach to patients with interactive voice recognition (IVR) to patients are promising interventions to overcome the barriers that physicians and patients encounter in treating hypertension and hyperlipidemia. While recent studies have begun to demonstrate the effectiveness of CDS in the ambulatory setting, there is an urgent need to implement and evaluate these systems in the practices of physicians practicing solo or in small groups in the community, outside the extensive HIT infrastructure of academic medical centers and integrated delivery systems.

IVR is a patient-outreach intervention that involves automated telephone calls to patients to patients in a conversation about specific health-related issues. Randomized control trials (RCTs) have shown that IVR monitoring with clinician follow-up can improve self-care, perceived health status, and physiologic outcomes among individuals with diabetes and hypertension.

The specific aim of this project is to evaluate, the effectiveness of CDS alone compared to IVR to improve the use of antihypertensive and lipid-lowering medications in community-based primary care practices.

ELIGIBILITY:
Inclusion Criteria:

* MDs, NPs, PAs, or DOs practicing in primary care or medical subspecialties and using eClinical Works EHR
* Patients of eligible physicians who have hypertension or hyperlipidemia

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
The main outcome measure will be the proportion of patients at treatment goal. | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Simon, MD, MPH, Principal Investigator — Brigham and Women's Hospital; David W Bates, MD, MSc, Principal Investigator — Brigham and Women's Hospital